CLINICAL TRIAL: NCT04018651
Title: Optimizing PrEP Utilization Among Alcohol and Other Drug (AOD) Using Women of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, jessy g devieux, Principal Investigator, Florida International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIU IRB 105978
Record Dates: First submitted 2019-06-17; First posted 2019-07-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: HIV Prevention
Keywords: Pre-Exposure Prophylaxis; PrEP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP Master Adherence Intervention (Experimental): The intervention consists of an introductory session and 4 individual sessions led by the PrEP Master, over an 8 week period. Between the sessions, the PrEP Master will conduct weekly check-in calls to participants to encourage adherence and assist with difficulties. During the weekly check-in, side effects and their impact will be assessed using assessment measures.
  Interventions: Behavioral: PrEP Master Adherence Intervention

INTERVENTIONS:
Behavioral: PrEP Master Adherence Intervention — The PrEP Master Adherence Intervention consists of 4 face to face individual education sessions and a series of telephone contacts to identify barriers and facilitators to optimal PrEP adherence over a six-month period. Each PrEP Master education session includes a review of an individualized plan to reduce risk, review of information about PrEP, and different discussion points. Key messages include:
  1. Importance of daily adherence;
  2. Three week delay for full effectiveness describing PrEP like taking the birth control pill;
  3. Condom use for other sexually transmitted infection (STI) prevention;
  4. Pregnancy prevention plans;
  5. Plans for follow up calls
  6. Referral to other treatment services if necessary

SUMMARY:
Nationally, the HIV case rate among black/ African American (AA) women is nearly 20 times higher than in white women; for Hispanic/Latino women it is 4.5 times higher. Moreover, according to findings in the HIV Prevention Trials Network (HPTN) Study 064 (The Women's HIV SeroIncidence Study), HIV incidence among women who live in communities with high HIV prevalence and poverty is about 6 times higher than for black/AA women. South Florida's new HIV diagnoses are now triple the national average due to rates in Miami-Dade and Broward counties in its AA, Latino and Haitian communities. Black women follow black men who have sex with men (MSM) as the most crisis-ridden of the communities in South Florida, the state as a whole, the South, and the U.S. Women overall have been at a disadvantage in the HIV epidemic due to gender differences and norms that shape biological, social and economic vulnerability. Racial and ethnic disparities magnify the risk. Co-factors such as alcohol and other drug (AOD) use intersect and reinforce other comorbidities. Living in a high prevalence area significantly hardens the risk and makes it tougher to overcome. Options to help women stay HIV negative have been limited, and the absence of practical female-controlled prevention strategies and relative dependence on cooperative use of the male condom continue to keep women's HIV vulnerability high. This obstacle shifted several years ago with FDA approval and Centers for Disease Control and Prevention's (CDC) endorsement of oral pre-exposure prophylaxis (PrEP). However, women do not know about PrEP. Despite FDA approval in 2012, followed by expansions in recommended use from the CDC and World Health Organization (WHO), the majority of women in the U.S. are not aware of oral PrEP as an HIV prevention strategy that applies to them. This study utilizes community-based participatory research (CBPR) to develop an intervention program that will promote optimal PrEP utilization among women of color in South Florida. The overall goal is to determine how best to target and improve PrEP utilization among women of color with substantial risks for HIV, including alcohol use.

DETAILED DESCRIPTION:
A singular limitation in the fight against HIV has been the absence of practical female-controlled prevention strategies and relative dependence on cooperative use of the male condom. Since 2012, medication for pre-exposure prophylaxis or PrEP has been FDA-approved in the U.S., with guidance for its use extended to all individuals at substantial risk in 2014 by the CDC and in 2015 by the WHO. In June 2016, the American Medical Association (AMA) instituted policies in concurrence, and in July 2016 an updated National HIV/AIDS Strategy was released making PrEP one of the four pillars in the nation's effort against HIV. To date, the largest uptake and implementation has been among the MSM population, which still bears the primary burden of the epidemic in the U.S. However, women continue to face a highly disproportionate risk and significant barriers to progress due to gender and structural disparities and biological susceptibility. Many of these barriers revolve around disparities that limit agency, most pointedly in negotiation of safe sex. Yet, existing studies indicate that very few of the women at substantial risk in the U.S. have awareness of PrEP, either from community sources or their doctors. Moreover, a recent national survey showed that PrEP awareness is suboptimal among a majority of providers. Clearly, PrEP as a viable female-controlled method is a long way from being a key part of the country's HIV strategy, and will require a community-driven approach to address demand and supply, uptake and accessibility, to shift the terms of women's agency in HIV prevention. This need is greatest among women of color, particularly when the use of alcohol and other drugs (AOD) severely compounds their risk.

This U34 utilizes community-based participatory research (CBPR) to build upon a Pre-Meeting of Community Stakeholders from the greater Miami and Fort Lauderdale areas, to develop an intervention program that will promote optimal PrEP utilization among women of color in South Florida who engage in risky sex and alcohol use. What is most potent in a CBPR-based study, is community participation in defining problems and intervention components, identifying applicable theories and evidence-based interventions (EBIs), and interpreting data and outcomes. The research team is currently conducting an exploratory pilot test in Miami-Dade County in South Florida, which leads the state in new HIV infections, and has a large multiethnic distribution of Black and Latino women in its population. Florida currently ranks 1st in HIV diagnoses among all states in the U.S. The overall goal is to determine how best to target and improve PrEP utilization among women of color with substantial risks for HIV, including alcohol use.

The investigator's Specific Aims are:

Aim 1: Identify perceived needs, priorities, barriers, and community strengths in the implementation of HIV prevention programs, with the development of a PrEP continuum care model, by conducting a summit to engage a diverse range of HIV- and HIV+ women of color, health care providers and community stakeholders.

Aim 2: Produce a replicable implementation program, including manuals, materials, screening and assessment instruments, and procedures, through the formation of a Community Advisory and Advocacy Board (CAAB) from summit participants, who will participate in a 2-day orientation training workshop and form working groups with research team members to formulate study methods and the intervention model.

Aim 3: Conduct an exploratory pilot of the PrEP model, implemented by the CAAB, in Broward and Miami-Dade for fidelity, feasibility, and acceptability, among 120 multi-ethnic women of color in South Florida (primarily African American (AA), Latina, Haitian). PrEP uptake and adherence and retention in care will be measured over a 6 month period. Results will inform a future U01, including the design of target and comparison groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 + years of age;
* born female;
* Identifies as female;
* Identifies as African American, Hispanic/Latina or Haitian (self or parent);
* Able to provide informed consent;
* HIV uninfected;
* Sexual risk (previous STI, inconsistent condom use, transactional sex, HIV infected partner);
* History of alcohol or drug use in last 3 months;
* No uncleared PrEP contraindications;
* No psychosis.

Exclusion Criteria:

* Less than 18 years of age
* male gender assignment at birth
* current male gender identity
* does not identify as African American, Haitian or Hispanic/Latina (self or parent)
* reports history of or current untreated psychosis
* unable to provide informed consent
* HIV infected
* Refuses PrEP medication
* Untreated medical contraindication for PrEP

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender identity
Enrollment: 38 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants receiving 3 Medication Appointments | 3 months
  Number of Participants who receive 3 refills of medication for PrEP
Percentage Adherence to PrEP Medication | 3 months
  Percentage adherence based on Pill count of remaining prescription medication at 3 months
Self reported PrEP Adherence | 3 months
  Percentage Adherence to daily PrEP medication via self report at 3 months
Number of Participants reporting Adherence to HIV testing recommendation | 3 months
  Number of Participants Receiving HIV test at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessy G Dévieux, Ph.D., Principal Investigator — Florida International Univ.
Locations (1):
- Florida International University Biscayne Bay Campus, North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No